CLINICAL TRIAL: NCT06503367
Title: Establishing Clinical Trial Readiness for Children 0-5 Years With Congenital Muscular Dystrophy Secondary to LAMA2 Mutations (READY CMD LAMA2)
Brief Title: Observation Study in Patients Age 0-5 Years With LAMA2-related Congenital Muscular Dystrophy
Status: Recruiting | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Iowa (Other); Washington University School of Medicine (Other); Stanford University (Other); University of Utah (Other); University of Rochester (Other); University of Pittsburgh (Other); University of Texas, Southwestern Medical Center at Dallas (Other); University of Minnesota (Other); University of California, Los Angeles (Other); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Anne M. Connolly, Principle Investigator, Nationwide Children's Hospital
Other Study IDs: Ready CMD LAMA2; 1U01NS124961-01A1 (NIH)
Record Dates: First submitted 2024-06-21; First posted 2024-07-16 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-02

CONDITIONS: LAMA2-MD (Merosin Deficient Congenital Muscular Dystrophy, MDC1A)
Keywords: Early Phase 1; Observational; Natural History; Neuromuscular; Functional Assessments
MeSH Terms: conditions — Muscular dystrophy congenital, merosin negative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to understand how young children with LAMA2-related dystrophy move and change over time. We will also learn about how this condition impacts other body systems.

Participants will undergo:

* Neuromuscular assessments
* Blood collections
* Swallowing and breathing assessments
* Questionnaires

DETAILED DESCRIPTION:
READY CMD LAMA2 is a Pre-Phase 1, single-arm, multicenter, prospective natural history clinical study to evaluate the natural history and potential early outcome measures in subjects with laminin α2-related dystrophy (LAMA2-RD) aged 0-5 years. The study seeks to enroll 44 subjects across 14 sites. NCH will enroll 10 subjects.

Subjects will complete in-person visits at Baseline, Month 6, Month 12, Month 18, and Month 24. Within two weeks of the Baseline, Month 12, and Month 24 visits, a remote visit will be performed to repeat and compare remote outcomes with in-person outcomes. Remote visits only will also be performed at Month 3 and Month 9. Adverse events will be captured every three months, beginning at baseline. Phone calls will be made by the coordinator and/or other delegated study staff at months 3, 9, 15, and 21.

The total study duration for each subject is up to 24 months.

Physical assessments to be performed will depend on the subject's age and may include the following:

* Assessment of motor milestones (maintained, lost or acquired)
* Neuromuscular Gross Motor Outcome (GRO)
* Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP-INTEND)
* Motor Function Measure (MFM-20)
* Bayley-4
* Respiratory assessments: capnography and collection of data on use of non- invasive ventilation and other respiratory support
* Physical exam
* Swallow/oromotor assessment: To be performed by physician, occupational therapist, speech language pathologist, or other licensed professional at the site.
* Muscle ultrasound may be performed at some sites.

Other assessments:

* Growth parameters [head circumference, chest circumference, length, weight, body mass index (BMI)]
* 12-lead electrocardiogram
* Mode of feeding
* Peds Quality of Life (PedsQL) Neuromuscular Module
* Pediatric Evaluation of Disability Inventory (PEDI)
* Clinical Global Impression of Change (CGIC), physician and parent/caregiver assessed.
* Blood samples will be collected from subjects and stored for biomarker and other research purposes. Blood samples will be collected at each in-person visit.
* Data from electronic medical records of evaluations performed as standard of care visits will be collected.

Medical history, concomitant medications, and AEs will be collected and assessed for a potential relationship to participation in this study.

The total duration of the study for each subject is up to approximately 24 months. A subject will be considered to have competed the study if he/she has completed all assessments up to and including Month 24 assessments. The end of the study is defined as the date of completion of the last scheduled assessment shown in the Schedule of Events for the last subject in the study.

Subjects who prematurely discontinue study participation will be encouraged to complete an End-of- Study Visit to include assessment of motor milestones and recording of AEs.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by the subject, parent(s) or legally authorized representative (LAR) and/or assent by the subject (when applicable).
* Subject must be aged birth to less than 5.0 years of age at time of consent.
* A confirmed diagnosis of LAMA2-RD confirmed via:

  a: Two pathogenic variants in the LAMA2 gene (via a CLIA-approved laboratory) or: b. muscle biopsy with absence of merosin (laminin-211) and at least one pathogenic variant in the LAMA2 gene
* Absence of another confirmed genetic disease.
* Willingness to maintain current exercise and/or physical therapy regimen for the duration of the clinical study.
* Willingness to comply with the study protocol, including but not limited to, all study procedures and visits.

Exclusion Criteria:

* Acute medical illness or hospitalization within 30 days prior to informed consent.
* Participation in a previous trial of any investigational agent for LAMA2-RD within 1 month prior to informed consent, or use of any other investigational therapy (including off-label use of Losartan) within 30 days prior to informed consent, or participation in other clinical studies, within 30 days (or 3 half-lives, whichever is longer) prior to informed consent, which in the opinion of the PI, may potentially confound results from this study.
* Other significant medical condition, which in the opinion of the site Principal Investigator may confound interpretation of the clinical course of LAMA2- RD.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study population will be neuromuscular clinic patients of site principal investigators, as well as individuals identified by our genetic counselor.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Validate the change over 24 months using the Neuromuscular Gross Motor Outcome | 24 months
  The Neuromuscular GRO is a 50-item assessment that measures a child's gross motor function when lying down, sitting, crawling, walking, jumping, and climbing stairs.
Validate the change over 24 months using the Bayley Scales of Infant and Toddler Development™ 4th Ed (BayleyTM-4) | 24 months
  The Bayley assess four areas of development: Gross Motor, Fine Motor, Speech and Language, and Social. These results are compared to typically developing children ages 15 days to 42 months. The entire assessment takes between 1 and 3 hours, with breaks.
Validate the change over 24 months using the Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders | 24 months
  The CHOP-Intend includes 16-items to measure a child's ability to move their body in a lying down position, supported sitting, and assisted rolling.
Validate the change over 24 months using the Motor Function Measure Scale-Short Form | 24 months
  The MFM-20 contains 20 items to assess a child's motor function in sitting, lying down, standing, and completing tabletop activities.
Validate the change over 24 months using the World Health Organization motor milestones | 24 months
  A child will be asked to complete 6 items to assess attainment of gross motor milestones including sitting without support, crawling, standing, and walking with and without assistance.

OTHER OUTCOMES:
Validate CK Biomarkers | From enrollment to the end of observation at 2 years.
  Blood will be drawn at each in-person visit to test Creatine Kinase, a muscle enzyme, and to store biomarkers for future research.
Muscle Ultrasound | 24 months
  Biceps or Quadriceps thickness will be measured in the middle of the muscle using standard ultrasound guidance.

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Connolly, MD, Principal Investigator — Nationwide Childrens Hospital
Locations (14):
- United States (14):
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - National Institute of Neurological Disorders and Stroke, NIH, Bethesda, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota, Saint Paul, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah